CLINICAL TRIAL: NCT06666205
Title: Evaluation of the Effect of Carbohydrate Quality on Sleep Quality and Depression in Patients with Type 2 Diabete
Brief Title: Carbohydrate Quality and Its Impact on Sleep and Depression in Type 2 Diabetes
Status: Completed | Type: Observational
Sponsor: Ankara Yildirim Beyazıt University (Other)
Responsible Party: Principal Investigator, Emine Elibol, Assist. Prof., Ankara Yildirim Beyazıt University
Other Study IDs: AYBUELİBOL002
Record Dates: First submitted 2024-10-22; First posted 2024-10-30 (Actual); Last update posted 2024-11-20 (Actual); Status verified 2024-10

CONDITIONS: Type 2 DM
Keywords: carbohydrate quality; type 2 diabetes mellitus; sleep quality; depression; stress
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Sleep Initiation and Maintenance Disorders; Depression

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Type 2 DM patients: This study focuses on patients with Type 2 diabetes and examines the impact of carbohydrate quality on sleep quality and depression. Participants were assessed using a demographic questionnaire, and their dietary carbohydrate intake was analyzed. Sleep patterns were monitored, and depression levels were measured using validated assessment scales. The study aims to investigate the relationship between carbohydrate quality, sleep health, and depression in this population.

SUMMARY:
The aim of this study was to evaluate the effect of carbohydrate quality on sleep quality and depression in patients with Type 2 diabetes. Data were collected from 150 patients with Type 2 diabetes mellitus using a demographic structure questionnaire, the Sleep Quality Scale (SQS), the Depression, Anxiety, and Stress Scale (DASS), and a Food Consumption Frequency Form. The data were analyzed using SPSS 26.

DETAILED DESCRIPTION:
Objective: The aim of this study was to evaluate the effect of carbohydrate quality on sleep quality and depression in patients with Type 2 diabetes.

Method: A total of 150 individuals with Type 2 diabetes were included in the study. A demographic questionnaire, the Sleep Quality Scale (SQS) (where a higher SQS score indicates lower sleep quality), and the Depression Anxiety and Stress Scale were administered to the participants. Additionally, data on the frequency of food consumption for 132 foods were obtained from the participants. To determine the Carbohydrate Quality Index (CQI) score, each of these four components (fiber intake, whole grain ratio, glycemic index, and total carbohydrate ratio) was evaluated on a scale of 1 to 5 points. The score for each component was then calculated, with Q5 indicating the best and Q1 indicating the worst carbohydrate quality. The data were analyzed using SPSS 24 software.

Detailed Description: This study will evaluate carbohydrate quality index ranges (Q1-Q5), sleep quality scale score, depression, stress, anxiety score, body mass index, diabetic age, sleep duration, body weight, daily macro and micro nutrients.

Conclusion: Results will be analyzed and interpreted after data collection is completed, and conclusions will be drawn accordingly.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 19 to 64 years
* Diagnosed with Type 2 diabetes mellitus
* Voluntary participation

Exclusion Criteria:

* Patients with cancer
* Pregnant and lactating women
* Individuals with alcohol or drug addiction
* Individuals diagnosed with psychiatric or neurological disorders

Ages: 19 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Community sample in Ankara, Turkey
Sampling Method: Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2023-04-01 (Actual); Primary Completion 2024-02-25 (Actual); Study Completion 2024-06-15 (Actual)

PRIMARY OUTCOMES:
Evaluating carbohydrate quality | Baseline
  A total of 132 food groups obtained from the food consumption frequency questionnaire were analyzed. Intake (g/day) was calculated using the BeBiS program with a global database, taking into account the amount and frequency of food consumed by each participant. Glycemic Index (GI) values were determined using the BeBiS program's global nutrient database, considering the amount and frequency of food consumed by each participant. To determine the Carbohydrate Quality Index (CQI) score, each of these four components (fiber intake, whole grain ratio, glycemic index, and total carbohydrate ratio) was evaluated on a scale of 1 to 5 points. The scores for each component were then calculated, with Q5 indicating the best and Q1 indicating the worst carbohydrate quality.

SECONDARY OUTCOMES:
Calculating sleep quality | Baseline
  The Sleep Quality Scale (SQS) was used to evaluate the sleep quality of individuals diagnosed with Type 2 diabetes mellitus. The scale consists of a total of 8 questions, each with 3 response options. Scores can range from a minimum of 7 to a maximum of 21. As the score obtained from the scale increases, sleep quality decreases. Questions 5 and 6 were reverse-scored, and a total score was calculated.
Depression, anxiety and stress scores | Baseline
  The Depression Scale was used to evaluate the psychological status of patients with Type 2 diabetes during this process. The scale consists of a total of 21 questions, each graded on a scale from normal to very advanced (mild, moderate, severe, advanced). It has three sub-dimensions: depression, anxiety, and stress. As the scores in the subscales increase, levels of depression, anxiety, and stress also increase.
Sociodemographic characteristics (age,) | Baseline
  Sociodemographic characteristics will be assessed using a structured questionnaire developed by the researchers. The questionnaire will include items measuring age, gender, education level, and income status. The results will be presented as numbers and percentages for each characteristic
Body Mass Index (BMI) | Baseline
  Kilograms per square meter (kg/m2)
Body weight | Baseline
  Body weight in kg
Height | Baseline
  Height in cm

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara Yıldırım Beyazıt University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No